CLINICAL TRIAL: NCT07183085
Title: Digital Care Programs for Mental Health: a Large-scale, Multi-disorder, Observational Study
Brief Title: Digital Care Programs for Mental Health
Status: Enrolling by invitation | Type: Observational
Sponsor: Sword Health, SA (Industry)
Responsible Party: Sponsor
Other Study IDs: SH-OBS-MND-US-01
Record Dates: First submitted 2025-09-10; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Mental Distress; Mental Resilience
MeSH Terms: interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: This program is designed to support individuals experiencing mental distress to improve overall wellbeing and mood symptom improvement.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Digital mental health program incorporating personalized physical and mental health exercises focused on physical activity, sleep hygiene, and mindfulness.

SUMMARY:
The purpose of this study is to create a research repository, composed of data collected over the course of digital care programs for mental health distress delivered by Sword Mind to individuals.

This will allow the investigators to observe the acceptance, engagement, and outcomes of programs using this approach in the treatment of multiple mental health concerns.

DETAILED DESCRIPTION:
Purpose This patient registry was designed as a research repository, composed of data collected over the course of digital care programs for mental health distress delivered by Sword Mind to individuals.

This data will allow the researchers to:

1. Assess the adoption, engagement and feasibility of digital care programs for mental distress;
2. Assess the results of digital care programs and compare the costs with the benefits obtained;
3. Correlate the results with participant's demographic and clinical profiles;
4. Examine the impact of mental health and the behavioral modification components of Mind's interventions on disease markers, comorbidities, and productivity;
5. Increase the knowledge on mental distress, namely how mental health distress symptoms progress and respond to digital care programs;
6. Develop new or improved tools to assist clinicians in the management of these disorders and in helping people achieve better mental health.

Design Prospective, observational

Participants This program is designed to support individuals experiencing mental distress to improve overall wellbeing and mood symptom improvement.

Participants will have access to a digital mental health program incorporating personalized physical and mental health exercises focused on physical activity, sleep hygiene, and mindfulness

Outcomes The primary outcome will be the evolution of the participant's mental health condition along the program. Depending on the condition, primary and secondary outcome measures vary, but the registry will include, in all cases, a complete characterization of the participant's mental health status, as well as the periodic assessment of: a) performance indicators (through condition-specific tests); b) patient-reported outcomes (obtained using internationally validated pathology-specific questionnaires); c) compliance; d) patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above;
* able to understand study procedures and willing to provide informed consent.

Exclusion Criteria:

* suicidal ideation with plan in the past 6 months;
* self-reported scores of the Patient Health questionnaire-9 (PHQ-9) above 19;
* suffering from any of the following mental health conditions: Schizophrenia, Bipolar Disorder, Alcohol Use Disorder, Substance Use Disorder, Eating Disorder, Post-Traumatic Stress Disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This program is designed to support individuals experiencing mental distress to improve overall wellbeing and mood symptom improvement.
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2035-09 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Assessed at baseline (upon initiation of the program) and then at regular intervals (5, 9, 15, 21, and 27 days). Additional follow-up assessments may be undertaken at other follow-up times: 3 months, 6 months and 12 months.
  Measured through the General Anxiety Disorder-7 (GAD-7), a 7-item scale (scores 0-21). Higher scores mean higher anxiety levels.
Depression | Assessed at baseline (upon initiation of the program) and then at regular intervals (5, 9, 15, 21, and 27 days). Additional follow-up assessments may be undertaken at other follow-up times: 3 months, 6 months and 12 months.
  Measured through the Patient Health Questionnaire-9 (PHQ-9), a 9-item scale (scores 0-27). Higher scores mean higher depression levels.

SECONDARY OUTCOMES:
Overall Improvement (PGIC) | Assessed at regular intervals (5, 9, 15, 21, and 27 days). Additional follow-up assessments may be undertaken at other follow-up times: 3 months, 6 months and 12 months.
  Measured through the Patient Global Impression of Change (PGIC) questionnaire. Scores reflect the participant's perceived overall improvement (range 1-7), with higher scores indicating greater improvement.
Self-reported Quality of Life | Assessed at baseline (upon initiation of the program) and then at regular intervals (5, 9, 15, 21, and 27 days). Additional follow-up assessments may be undertaken at other follow-up times: 3 months, 6 months and 12 months.
  Assessed through the question "On a scale of 0-100, how would you rate your overall health, with 0 being the worst health imaginable and 100 the best health imaginable?"
Work productivity and absenteeism | Assessed at baseline (upon initiation of the program) and then at regular intervals (5, 9, 15, 21, and 27 days). Additional follow-up assessments may be undertaken at other follow-up times: 3 months, 6 months and 12 months.
  Measured through Work Productivity and Activity Impairment Questionnaire (WPAI) assessed by the sub-scores: WPAI overall (combining presenteeism and absenteeism), WPAI work (presenteeism), WPAI time (absenteeism) and WPAI activities (activities of daily living impairment) (scores 0-100%). Higher scores mean greater impairment.
Sleep Duration (wearable-measured) | Recorded daily. Outcomes summarized at regular intervals (5, 9, 15, 21, and 27 days). Additional follow-up assessments may be undertaken at other follow-up times: 3 months, 6 months and 12 months.
  Sleep will be assessed using a wearable device, including the total number of hours spent sleeping.

OTHER OUTCOMES:
Program Activities Performed | through study completion, an average of 3 months
  Number of total activities performed, including those related to the mindfulness, physical activity, or sleep-related components.
Total Program Activities Time | through study completion, an average of 3 months
  Number of minutes spent on activities (aggregated), including those related to the mindfulness, physical activity, or sleep-related components.
Self-reported satisfaction | Assessed at regular intervals (5, 9, 15, 21, and 27 days). Additional follow-up assessments may be undertaken at other follow-up times: 3 months, 6 months and 12 months.
  Measured through the Net Promoter Score question collected at end of program: "On a scale from 0 to 10, how likely are you to recommend SWORD's programs to a friend or family member?")
Average Program Activities Time per Week | through study completion, an average of 3 months
  Average number of minutes spent on program activities per week, including those related to the mindfulness, physical activity, or sleep-related components.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando D Correia, MD, PhD, Principal Investigator — SWORD HEALTH INC
Locations (1):
- Sword Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No